CLINICAL TRIAL: NCT04995510
Title: Examination of Respiratory Muscle Function, Diaphragm Thickness and Health Related Physical Fitness Parameters in Chronic Obstructive Pulmonary Disease Individuals
Brief Title: Respiratory Muscle Function, Diaphragm Thickness and Health Related Physical Fitness Parameters in Individuals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Eylem TÜTÜN YÜMİN, Associate Professor, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-ETY-01
Record Dates: First submitted 2021-07-10; First posted 2021-08-09 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; diaphragm thickness; respiratory muscle function; body composition; physical fitness
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Obstructive Pulmonary Disease Group: Individuals diagnosed with chronic obstructive pulmonary disease by ''Bolu Abant Izzet Baysal University'' Faculty of Medicine, Department of Chest Diseases and referred to the Physiotherapy and Rehabilitation Department of Bolu Abant Izzet Baysal University Health Sciences Faculty
  Interventions: Other: Observational
- Healthy Group: Volunteer healthy individuals with similar demographic characteristics and without any diagnosed disease will be recruited
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — To evaluate your chronic obstructive pulmonary disease with Chronic Obstructive Pulmonary Disease assessment test, respiratory muscle strength with intraoral pressure measurement device, respiratory muscle endurance with increasing threshold load respiratory muscle endurance test, diaphragm thickness with ultrasound device, cardiorespiratory fitness with 6 Minute Walk Test, flexibility trunk lateral flexion test , back scratch test and sit and lie down test, muscle strength and endurance will be evaluated with push-up test, sit-up test, sit and stand test and hand grip strength, body composition will be evaluated by bioelectrical impedance analysis, physical activity will be questioned with the International Physical Activity Assessment Questionnaire, shortness of breath with the Mmrc Dyspnea Scale, and perception of fatigue and shortness of breath with the Modified Borg Scale.

SUMMARY:
In the literature, studies evaluating respiratory muscle function, diaphragm thickness and health-related physical fitness parameters together are insufficient in individuals with chronic obstructive pulmonary disease. In the thesis study, it is thought that the respiratory muscle function, diaphragm thickness, health-related physical fitness parameters, physical activity and lung functions of individuals with chronic obstructive pulmonary disease can be evaluated together to contribute to the literature. The aim of this study is to evaluate diaphragm thickness, respiratory muscle strength, endurance, body composition, aerobic exercise capacity, upper and lower extremity muscle strength and endurance, grip strength, flexibility in individuals with chronic obstructive pulmonary disease and compare them with the healthy group.

DETAILED DESCRIPTION:
Breathing is the exchange of oxygen and carbon dioxide gases with inspiration (breathing in) and expiration (breathing) in order to maintain the optimum oxygen level in arterial blood. Respiration takes place through respiratory muscles. While inspiration takes place through the diaphragm and accessory respiratory muscles; Expiration takes place passively. Respiratory muscle function is determined by evaluating respiratory muscle strength and respiratory muscle endurance together. respiratory muscle dysfunction; It is a decrease in respiratory muscle strength, endurance, or both, caused by factors such as elongated diaphragm fibers, increased respiratory workload, changes in muscle mass and abdominal weight. Today, respiratory muscle strength are widely used in the evaluation of respiratory muscle function. However, evaluation of respiratory muscle endurance is more effective than respiratory muscle strength in the evaluation of submaximal respiratory muscle contraction, which is valid for daily activities, and in the clinical, functional and prognostic evaluation of respiratory muscles. In chronic obstructive pulmonary disease, respiratory muscle function is associated with pulmonary functions, symptoms, comorbidities, health status, airway obstruction, lung volumes, and physiological disorders. Respiratory muscle dysfunction in chronic obstructive pulmonary disease increases with disease progression. Dysfunction in the diaphragm, which is the most important respiratory muscle, can be evaluated with respiratory muscle strength and endurance, as well as diaphragm thickness. Diaphragm thickness provides information about disease progression in individuals with chronic obstructive pulmonary disease. It is known that diaphragm thickness is associated with respiratory muscle strength and respiratory function parameters in individuals with chronic obstructive pulmonary disease.

The World Health Organization defines health as "a state of complete physical, social and mental well-being and not merely the absence of disease or infirmity". One of the important factors for maintaining health is physical fitness. physical fitness; It is the ability to perform occupational, recreational and daily activities correctly and successfully without fatigue. Physical fitness is also known as the ability to do daily tasks vigorously and carefully, without excessive fatigue, and to allocate sufficient energy for leisure and unexpected emergencies. Physical fitness is divided into two as health-related physical fitness and sports-related physical fitness. While health-related physical fitness parameters are body composition, cardiorespiratory fitness, muscular strength and endurance, flexibility; Sport-related physical fitness parameters are balance, coordination, reaction time, agility, speed and power. Decreased physical fitness in individuals with chronic obstructive pulmonary disease is associated with respiratory problems (such as airway obstruction). It is known that physical fitness is related to the ability to perform physical activity. Low physical fitness occurs in most individuals with chronic obstructive pulmonary disease due to decreased physical activity. There is an important relationship between physical fitness and lung functions.

In the literature, studies evaluating respiratory muscle function, diaphragm thickness and health-related physical fitness parameters together are insufficient in individuals with chronic obstructive pulmonary disease. In the thesis study, which is planned to be done, it is thought that the respiratory muscle function, diaphragm thickness, health-related physical fitness parameters, physical activity and lung functions of individuals with chronic obstructive pulmonary disease can be evaluated together to contribute to the literature.

The aim of this study is to evaluate diaphragm thickness, respiratory muscle strength, endurance, body composition, aerobic exercise capacity, upper and lower extremity muscle strength and endurance, grip strength, flexibility in individuals with chronic obstructive pulmonary disease and compare them with the healthy group.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with chronic obstructive pulmonary disease
* Be between the ages of 40-65
* No medication changes due to acute exacerbation for at least three weeks
* Be stable
* Volunteering to participate in research
* To cooperate
* Patients with written consent form
* Healthy individuals in a similar age range without a diagnosed disease and symptoms will be included

Exclusion Criteria:

* Those with a history of chronic obstructive pulmonary disease exacerbations
* Individuals with orthopedic disease
* Individuals with neurological disease
* Individuals with other co-existing lung and systemic diseases other than chronic obstructive pulmonary disease
* Those who have had major surgery in the past few months
* Individuals with a history of recurrent significant clinical infections
* Have cognitive problems
* Having had unstable angina,
* Previous Myocardial Infarction
* Individuals with severe congestive heart failure refractory to medical therapy, individuals with uncontrolled hypertension
* Individuals with cancer

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Obstructive Pulmonary Disease (COPD) is a common, preventable, and treatable disease characterized by persistent airflow limitation, usually progressive, associated with an increased chronic inflammatory response of the airways and lung to noxious gases and particles. In addition, healthy individuals in a similar age range without a diagnosed disease and symptoms will be included in the study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-12-18 (Estimated)

PRIMARY OUTCOMES:
Diaphragm Thickness | 5 minutes
  Diaphragm thickness will be measured by ultrasound. Diaphragm thickness will be measured twice, when the person fully exhales and fully fills their lungs with air. Diaphragm thickness will be measured at the 8th or 9th intercostal space. Decreased diaphragm thickness indicate impaired respiratory muscle function; being in the normal range indicates good respiratory muscle function.
Diaphragm Mobility | 5 minutes
  Diaphragm mobility will be measured by ultrasound. Diaphragm mobility will be done by using the total amount of movement of the diaphragm until the individual breathes completely from the point of exhalation. Diaphragm mobility will be performed at the intersection of the medial axillary line and the costal line. Decreased diaphragm mobility indicate impaired respiratory muscle function; being in the normal range indicates good respiratory muscle function.

SECONDARY OUTCOMES:
Measurement of Maximal Inspiratory Pressure | 5 minutes
  Maximal Inspiratory Pressure will be measured with an intraoral pressure measuring device. Maximal Inspiratory Pressure reflects respiratory muscle strength. An increase in Maximal Inspiratory Pressure indicates high respiratory muscle strength; A low Maximal Inspiratory Pressure value indicates respiratory muscle weakness.
Incremental Threshold Load Endurance Test | 10 minutes
  Respiratory muscle endurance will be measured with an incremental threshold load respiratory muscle endurance test. The respiratory muscle endurance test will be performed using a respiratory muscle training device. Endurance test is performed by breathing rapidly and deeply against the respiratory muscle training device of the individual. The individual should continue the test as long as possible. A high respiratory muscle endurance score indicates good respiratory muscle function; A low score indicates respiratory muscle dysfunction.
Pulmonary Function Test | 5 minutes
  Pulmonary function test will be performed with a spirometer according to the criteria of the American Thoracic Society and the European Respiratory Society. While the decrease in pulmonary function test parameters shows worsening of lung functions; parameters in the normal range indicate good lung functions.
Six Minute Walk Test | 10 minutes
  The six minute walk test will be used to evaluate functional exercise capacity. The individual will be asked to walk as fast as possible throughout the test. High walking distance indicates good exercise capacity; A low walking distance indicates a decrease in exercise capacity.
Body Composition: Lean Body Mass Percentage | 2 minutes
  The lean body mass percentage of the individual will be determined by Bioelectrical Impedance Analysis. The measurement will be made by the individual standing on the device with bare feet and waiting. If the lean body mass percentage values are in the normal range, the body composition is normal; lean body mass percentage low values indicate deterioration of body composition.
International Physical Activity Assessment Questionnaire | 2 minutes
  Physical activity level will be assessed with the short form of the International Physical Activity Assessment Questionnaire. The short form of the International Physical Activity Assessment Questionnaire consists of seven questions. A high questionnaire score indicates a high level of physical activity; A low score indicates physical inactivity.
Chronic Obstructive Pulmonary Disease Assessment Test (CAT) | 2 minutes
  Chronic Obstructive Pulmonary Disease Assessment Test is an eight-item scale measuring health status in Chronic Obstructive Pulmonary Disease. This scale is used to determine the health status of individuals with Chronic Obstructive Pulmonary Disease all over the world. Each question is scored between 0-5 and a total score between 0 and 40 is given. A score of 0 represents the best and a score of 40 represents the worst state of health.
Modified Medical Research Council Dyspnea Scale | 2 minutes
  It is a 5-item scale scored between 0-4 for individuals' shortness of breath. Evaluates dyspnea and activity limitation in individuals with chronic obstructive pulmonary disease. An increase in the score indicates an increase in shortness of breath.
Modified Borg Scale (MBS) | 2 minutes
  In this scale, in which the perception of shortness of breath at rest and during exercise will be evaluated, scoring varies between 0-10 points, although high scores indicate high breathlessness and fatigue.
Trunk Lateral Flexion Test: | 1 minute
  Lateral flexion flexibility is measured with the trunk lateral flexion test. While standing, the arms are held in an upright position with the feet parallel to the body and feet shoulder-width apart. First of all, the distance between the point where the right 3rd finger tip is located and the point where the finger tip is located after right lateral flexion is checked. The distance between the start point and the end point is recorded. The test is repeated three times and the best measurement is recorded as the result. A high distance indicates good trunk flexibility; The low distance indicates that the trunk flexibility is insufficient.
Back Scratching Test | 1 minute
  In the back scratch test, the palmar side of the upper hand and the back of the lower hand should be placed on the back and the distance of the third fingers to each other should be recorded. The test is repeated three times and the best result is considered the test result. If the distance is too much, it shows that the flexibility is bad; A low distance indicates good flexibility.
Sit-Reach Test | 1 minute
  In the sit-reach test, individuals are seated on a flat surface and the individual's feet are made to rest flat on the test bench. Then, the individual is asked to reach forward as much as possible. The test result is obtained by measuring the distance between the tip of the third finger and the foot. During the test, the individual is expected to wait 2-3 seconds at the last point and the test is repeated 3 times to record the best result. A high distance indicates good flexibility; If the distance is low, it indicates that the flexibility is bad.
30 Second Modified Push Up Test | 1 minute
  A 30 second modified push up test will be used to evaluate the upper body muscle strength and endurance of individuals. The individual, whose hands and knees are in contact with the floor, and whose knees and elbows are flexed on the mat, is asked to push his body backwards by extending his elbows without disturbing the flexion of the knees. The number of correct movements in 30 seconds will be recorded as the test result. A high number indicates good upper extremity muscle strength and endurance; A low number indicates poor upper extremity muscle strength and endurance.
Sit Up Test | 1 minute
  The 30-second sit-up test will be used to evaluate the strength and endurance of the abdominal muscles of the individuals. Individuals are asked to lock their hands on the nape in supine, hip and knee flexion, with the plantar face of the foot on the ground (hooked position), and starting from this position, individuals are asked to flex their trunk as much as possible until the scapula is out of contact with the ground. The number of trunk flexions for 30 seconds is recorded. A high number indicates good trunk muscle strength and endurance; A low number indicates poor trunk muscle strength and endurance.
Sit to Stand Test | 1 minute
  Sit and stand test can be performed to evaluate lower extremity muscle strength and endurance. Individuals are asked to cross their arms over their shoulders and sit and stand up for 30 seconds, and the number of sitting and standing is recorded. A high number indicates good lower extremity muscle strength and endurance; A low number indicates poor lower extremity muscle strength and endurance.
Hand Grip Strength | 1 minute
  Hand grip dynamometer is used to measure hand grip strength. Measurements are made three times on the left and right sides of the individual in a sitting position, shoulder adduction, elbow 90° flexion, and forearm neutral position. A high value indicates that the hand grip strength is good; A low value indicates a low hand grip strength.

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant İzzet Baysal University Department of Physiotherapy and Rehabilitation, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No